CLINICAL TRIAL: NCT05554237
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, SINGLE AND MULTIPLE-DOSE STUDY TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-07612577 (PF-06264006 [CTB] + PF-07338233 [AVP]) IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn About the Study Medicine Called CTB+AVP in Healthy Adult People.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C4691001; 2021-005428-39 (EudraCT Number)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-06

CONDITIONS: Healthy
MeSH Terms: interventions — Ceftibuten

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant and investigator-blinded and sponsor-open design for Part-1 and Part-2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PF-07612577 (Experimental): Part-1: Dose 1, Dose 2, Dose 4, Dose 5 Part-2: Cohort 2-5
  Interventions: Drug: PF-07612577
- Placebo (Placebo Comparator): Part-1: Dose 1-5 Part-2: Cohort 2-4
  Interventions: Drug: Placebo
- PF-06264006 (Experimental): Part-1: Dose 3, Dose 5
  Interventions: Drug: PF-06264006

INTERVENTIONS:
Drug: Placebo — Placebo
  Other Names: Placebo comparator
  Arms: Placebo
Drug: PF-07612577 — PF-07612577
  Other Names: CTB+AVP
  Arms: PF-07612577
Drug: PF-06264006 — PF-06264006
  Other Names: ceftibuten (CTB)
  Arms: PF-06264006

SUMMARY:
The purpose of this clinical trial is to learn about the pharmacokinetics, safety and tolerability of various single- and multiple-doses of CTB+AVP in healthy adult participants. CTB+AVP is a study medicine that is being developed to treat people with complicated urinary tract infections.

This study is seeking healthy adult male and female participants, 18-60 years of age, with a body weight > 50 kg and a BMI of 17.5 to 30.5 kg/m2.

Participants in Part-1 of the study will receive increasing single doses of CTB and/or AVP. Participants in Part-2 will receive increasing multiple doses of CTB+AVP three times a day for 7 days. The study team will monitor how each participant is doing with the study treatments via close monitoring in an in-patient setting. Experiences of people receiving CTB+AVP will be compared to those of people who do not. This will help determine if CTB+AVP is safe and well-tolerated at each dose of the study medicine.

Participants will take part in this study for a maximum of 12 weeks for Part-1 (up to 4 weeks for screening, up to 3 weeks of taking study medicine and up to 5 weeks for safety follow-up visit) and for a maximum of 10 weeks for Part-2 (up to 4 weeks for screening, up to 1 week of taking study medicine and up to 5 weeks for safety follow-up visit). During the duration of the study, blood samples for study medicine levels, and various measures for monitoring safety such as blood samples for clinical laboratory measurements, electrocardiograms and vital sign measurements will be taken.

DETAILED DESCRIPTION:
This is a 2-part study in healthy male and female adult participants.

Part-1 is to evaluate safety, tolerability and pharmacokinetics (PK) of 3 planned and 2 optional doses in 8 participants, in a 5-period sequential single dose design.

Part-2 is to evaluate safety, tolerability and PK of 1 planned and 2 optional cohorts in 8 participants each, in a multiple dose sequential design, with 7 days of repeated every 8 hours (q8h) dosing in each cohort. In addition, 2 optional cohorts in 6 participants each of Japanese descent and Chinese descent will also receive multiple doses of CTB+AVP repeated every 8 hours (q8h) for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
2. For optional Japanese cohort only: Japanese participants who have 4 Japanese biologic grandparents who were born in Japan
3. For optional Chinese cohort only: Chinese participants who were born in mainland China, and both parents are of Chinese descent.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing)
2. Known allergy to the cephalosporin group of antibiotics
3. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed
4. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality [or other conditions or situations related to COVID-19 pandemic (eg, Contact with positive case, residence, or travel to an area with high incidence)] that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
5. A positive urine drug test
6. Positive test result for SARS-CoV-2 infection at the time of screening or Day -1

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4691001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 42 participants (8 in Part 1 and 34 in Part 2) were enrolled in the study. The study was conducted at 1 site in Belgium.
Groups:
- CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1): Healthy participants were administered a single oral dose of ceftibuten(CTB) 400 milligrams (mg) along with Avibactam Prodrug (AVP) 900 mg on Day 1 of Period 1 followed by a single oral dose of CTB 800 mg along with AVP 1350 mg on Day 1 of Period 2. Participants received a single oral dose of CTB 800 mg alone on Day 1 of Period 3 followed by CTB 1200 mg with AVP 1350 mg and placebo for CTB 1600 mg orally on Day 1 of Period 4 and 5 respectively. There was a washout period of minimum 3 days between doses.
- CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1): Healthy participants were administered a single oral dose of CTB 400 mg along with AVP 900 mg on Day 1 of Period 1 followed by a single oral dose of CTB 800 mg along with AVP 1350 mg on Day 1 of Period 2. Participants received a single oral dose of CTB 800 mg alone on Day 1 of Period 3 followed by a placebo of CTB 1200 mg along with AVP 1350 mg and CTB 1600 mg orally on Day 1 of Period 4 and 5 respectively. There was a washout period of minimum 3 days between doses.
- CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1): Healthy participants were administered a single oral dose of CTB 400 mg along with AVP 900 mg on Day 1 of Period 1 followed by a single oral dose of placebo for CTB 800 mg along with AVP 1350 mg on Day 1 of Period 2. Participants received a single oral dose of placebo for CTB 800 mg alone on Day 1 of Period 3 followed by CTB 1200 mg along with AVP 1350 mg and CTB 1600 mg orally on Day 1 of Period 4 and 5 respectively. There was a washout period of minimum 3 days between doses.
- Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1): Healthy participants were administered a single oral dose of placebo for CTB 400 mg along with AVP 900 mg on Day 1 of Period 1 followed by a single oral dose of CTB 800 mg along with AVP 1350 mg on Day 1 of Period 2. Participants received a single oral dose of CTB 800 mg alone on Day 1 of Period 3 followed by CTB 1200 mg along with AVP 1350 mg and CTB 1600 mg orally on Day 1 of Period 4 and 5 respectively. There was a washout period of minimum 3 days between doses.
- CTB 400 mg + AVP 1350 mg q8h (Part-2): Healthy participants were administered CTB 400 mg along with AVP 1350 mg once every 8 hours (q8h) in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2): Healthy participants were administered placebo for CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- CTB 800 mg + AVP 1350 mg q8h (Part-2): Healthy participants were administered CTB 800 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2): Healthy participants were administered placebo for CTB 800 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- CTB 400 mg + AVP 900 mg q8h (Part-2): Healthy participants were administered CTB 400 mg along with AVP 900 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2): Healthy participants were administered placebo for CTB 400 mg along with AVP 900 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2): Healthy Japanese participants were administered CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2): Healthy Japanese participants were administered placebo for CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2): Healthy Chinese participants were administered CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
- Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2): Healthy Chinese participants were administered placebo for CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
Period: Part 1: Period 1 Treatment (1 Day)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 1 Washout (3 Days)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2 Treatment (1 Day)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 2 Washout (3 Days)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 3 Treatment (1 Day)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 3 Washout (3 Days)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 4 Treatment (1 Day)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 4 Washout (3 Days)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Period 5 Treatment (1 Day)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (7 Days)
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Started | 0 (No participants were enrolled in Part 2.) | 0 (No participants were enrolled in Part 2.) | 0 (No participants were enrolled in Part 2.) | 0 (No participants were enrolled in Part 2.) | 6 (Participants enrolled in Part 2 of the study.) | 2 (Participants enrolled in Part 2 of the study.) | 6 (Participants enrolled in Part 2 of the study.) | 2 (Participants enrolled in Part 2 of the study.) | 6 (Participants enrolled in Part 2 of the study.) | 2 (Participants enrolled in Part 2 of the study.) | 5 (Participants enrolled in Part 2 of the study.) | 1 (Participants enrolled in Part 2 of the study.) | 3 (Participants enrolled in Part 2 of the study.) | 1 (Participants enrolled in Part 2 of the study.)
Completed | 0 | 0 | 0 | 0 | 4 | 2 | 6 | 2 | 6 | 1 | 5 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants randomly assigned to study intervention and who take at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | CTB400+AVP900mg/CTB 800+AVP1350 mg /CTB800mg/ CTB1200+AVP1350 mg/Placebo for CTB 1600mg(Part1) | CTB400+AVP900mg /CTB800+AVP1350mg /CTB 800mg/Placebo for CTB1200+AVP1350 mg /CTB1600 mg(Part1) | CTB400+AVP900mg/ Placebo for CTB800+AVP1350mg/ Placebo CTB800mg/ CTB1200+AVP1350mg/ CTB1600mg(Part1) | Placebo for CTB400+AVP900mg/ CTB 800+AVP1350mg/ CTB800mg/ CTB1200mg+AVP1350mg/ CTB1600mg(Part1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1 | 42
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 2 | 2 | 1 | 2 | 2 | 1 | 6 | 2 | 4 | 2 | 4 | 0 | 2 | 0 | 30
  45-64 Years | 0 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 10
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Male | 1 | 2 | 2 | 1 | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 0 | 2 | 0 | 37
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 2 | 2 | 6 | 2 | 4 | 2 | 6 | 2 | 0 | 0 | 0 | 0 | 30
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 3 | 0 | 9
  Not disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Cis-Ceftibuten (CTB): Part 1
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: Pharmacokinetic parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported for the given part of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- CTB 400 mg + AVP 900 mg (Part-1): Healthy participants were administered a single oral dose of CTB 400 mg along with a single oral dose of AVP 900 mg in any of the treatment periods.
- CTB 800 mg + AVP 1350 mg (Part-1): Healthy participants were administered a single oral dose of CTB 800 mg along with a single oral dose of AVP 1350 mg in any of the treatment periods.
- CTB 800 mg (Part-1): Healthy participants were administered a single oral dose of CTB 800 mg in any of the treatment periods.
- CTB 1200 mg + AVP 1350 mg (Part-1): Healthy participants were administered a single oral dose of CTB 1200 mg along with a single oral dose of AVP 1350 mg in any of the treatment periods.
- CTB 1600 mg (Part-1): Healthy participants were administered a single oral dose of CTB 1600 mg in any of the treatment periods.
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram per milliliter (ng/mL) | 18170 (24) | 25470 (18) | 30510 (16) | 27120 (12) | 44990 (25)
Statistical Analysis 1: Comparison: CTB 800 mg + AVP 1350 mg (Part-1) vs CTB 800 mg (Part-1); Test type: Other; Ratio of adjusted geometric means = 83.46, 90% CI 2-sided [74.67 to 93.29] — Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect (for CTB 800 mg + AVP 1350 mg versus CTB 800mg only)

2. Primary Outcome: Time for Cmax (Tmax) of CTB: Part 1
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours | 3.21 [2.12 to 4.05] | 4.03 [3.03 to 4.15] | 3.50 [1.50 to 4.02] | 5.05 [4.03 to 6.05] | 4.01 [2.02 to 4.10]

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of CTB: Part 1
Description: AUClast was determined using the linear/log trapezoidal method.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram*hours per milliliter | 94050 (18) | 154100 (14) | 171800 (15) | 183600 (15) | 319200 (24)
Statistical Analysis 1: Comparison: CTB 800 mg + AVP 1350 mg (Part-1) vs CTB 800 mg (Part-1); Test type: Other; Ratio of adjusted geometric means = 89.70, 90% CI 2-sided [87.24 to 92.23] — Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect (for CTB 800 mg + AVP 1350 mg versus CTB 800mg only

4. Primary Outcome: Dose-Normalized Cmax (Cmax[dn]) of CTB: Part 1
Description: Dose-normalized Cmax was determined as Cmax/Dose.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram per milliliter per milligram | 45.45 (24) | 31.83 (18) | 38.16 (16) | 22.61 (12) | 28.12 (25)

5. Primary Outcome: Dose-Normalized AUClast (AUClast[dn]) of CTB: Part 1
Description: AUClast(dn) was determined as AUClast/Dose.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter per milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram*hour/milliliter per milligram | 235.2 (18) | 192.9 (14) | 214.9 (15) | 152.9 (15) | 199.6 (24)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of CTB: Part 1
Description: AUCinf was calculated as AUClast + (Clast/kel), where Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram*hour per milliliter | 94730 (18) | 155800 (13) | 173200 (14) | 184900 (15) | 321900 (24)
Statistical Analysis 1: Comparison: CTB 800 mg + AVP 1350 mg (Part-1) vs CTB 800 mg (Part-1); Test type: Other; Ratio of adjusted geometric means = 89.91, 90% CI 2-sided [87.47 to 92.41] — [estimate comment as in outcome 3, analysis 1]

7. Primary Outcome: Dose-Normalized AUCinf (AUCinf[dn]) of CTB: Part 1
Description: AUCinf(dn) was calculated as AUCinf/Dose.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter per milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Nanogram*hour/milliliter per milligram | 236.9 (18) | 194.6 (13) | 216.7 (14) | 153.8 (15) | 200.9 (24)

8. Primary Outcome: Terminal Half-Life (t1/2) of CTB: Part 1
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Hours | 3.073 (0.54265) | 2.708 (0.57031) | 2.908 (0.53905) | 3.138 (0.27600) | 3.180 (0.28817)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F) of CTB: Part 1
Description: Vz/F was calculated as Dose/(AUCinf * kel) where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Liter | 18.44 (20) | 19.70 (14) | 19.10 (16) | 29.28 (14) | 22.72 (30)

10. Primary Outcome: Apparent Clearance (CL/F) of CTB: Part 1
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Liter per hour | 4.221 (18) | 5.136 (13) | 4.620 (14) | 6.492 (15) | 4.973 (24)

11. Primary Outcome: Maximum Observed Concentration (Cmax) of AVP, Avibactam (AVI) and Hydroxy Pivalic Acid (HPA): Part 1
Description: The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: Pharmacokinetic parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported for the given part of the study. Data is reported for CTB 400 mg + AVP 900 mg, CTB 800 mg + AVP 1350 mg and CTB 1200 mg + AVP 1350 mg arms only as only participants from these arms received AVP (AVI and HPA: metabolites of AVP).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter
  AVP | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI | 3856 (44) | 5955 (13) | 6714 (26)
  HPA | 1521 (33) | 2552 (14) | 2676 (36)

12. Primary Outcome: Dose-Normalized AUClast (AUClast[dn]) of AVP, AVI and HPA: Part 1
Description: AUClast(dn) was determined as AUClast/Dose. The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hour/milliliter/milligram
  AVP: number analyzed (Participants) | 6 | 6 | 5
  AVP | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI | 36.10 (33) | 40.91 (13) | 41.67 (19)
  HPA | 37.04 (24) | 43.89 (11) | 43.59 (23)

13. Primary Outcome: Time for Cmax (Tmax) of AVP, AVI and HPA: Part 1
Description: The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: Pharmacokinetic parameter analysis set. Data is reported for CTB 400 mg + AVP 900 mg, CTB 800 mg + AVP 1350 mg and CTB 1200 mg + AVP 1350 mg arms only as only participants from these arms received AVP (AVI and HPA: metabolites of AVP). Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Median (Full Range); unit: Hours
Groups:
- CTB 1200 mg + AVP 1350 mg (Part-1): Healthy participants were administered a single dose of CTB 1200 mg and AVP 1350 mg orally on day 1 in period 4
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  AVP: number analyzed (Participants) | 1 | 0 | 2
  AVP | NA [NA to NA] — Data could not be calculated as values were below limit of quantification. |  | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  AVI | 4.01 [2.08 to 6.00] | 3.50 [1.50 to 6.00] | 4.50 [2.50 to 6.02]
  HPA | 4.01 [1.50 to 6.00] | 4.00 [1.00 to 6.00] | 4.50 [2.50 to 6.02]

14. Primary Outcome: Dose-Normalized Cmax (Cmax[dn]) of AVP, AVI and HPA: Part 1
Description: Dose-normalized Cmax was determined as Cmax/Dose. The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter per milligram
  AVP | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI | 6.388 (44) | 6.583 (13) | 7.422 (26)
  HPA | 5.635 (33) | 6.300 (14) | 6.608 (36)

15. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of AVP, AVI and HPA: Part 1
Description: AUClast was determined using the linear/log trapezoidal method. The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hours per milliliter
  AVP: number analyzed (Participants) | 6 | 6 | 5
  AVP | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI | 21760 (33) | 37000 (13) | 37680 (19)
  HPA | 9996 (24) | 17790 (12) | 17670 (23)

16. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of AVP, AVI and HPA: Part 1
Description: as for outcome 6
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hours per milliliter
  AVP: number analyzed (Participants) | 0 | 0 | 0
  AVI | 22050 (34) | 38060 (13) | 38090 (19)
  HPA | 10220 (24) | 18440 (10) | 17950 (22)

17. Primary Outcome: Dose-Normalized AUCinf (AUCinf[dn]) of AVP, AVI and HPA: Part 1
Description: AUCinf(dn) was calculated as AUCinf/Dose.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hour/milliliter/milligram
  AVP: number analyzed (Participants) | 0 | 0 | 0
  AVI | 36.58 (34) | 42.10 (13) | 42.11 (19)
  HPA | 37.86 (24) | 45.59 (10) | 44.35 (22)

18. Primary Outcome: Terminal Half-Life (t1/2) of AVP, AVI and HPA: Part 1
Description: as for outcome 8
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  AVP: number analyzed (Participants) | 0 | 0 | 0
  AVI | 4.043 (1.0748) | 5.302 (1.4722) | 3.632 (0.86092)
  HPA | 4.218 (0.92090) | 5.347 (1.5405) | 3.853 (0.86710)

19. Primary Outcome: Apparent Volume of Distribution (Vz/F) of AVP, AVI and HPA : Part 1
Description: as for outcome 9
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Liter
  AVP: number analyzed (Participants) | 0 | 0 | 0
  AVI | 154.6 (27) | 175.0 (33) | 121.5 (33)
  HPA | 157.6 (24) | 163.2 (35) | 122.7 (36)

20. Primary Outcome: Apparent Clearance (CL/F) of AVP, AVI and HPA: Part 1
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,14 and 24 hours post dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1)
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour
  AVP: number analyzed (Participants) | 0 | 0 | 0
  AVI | 27.35 (34) | 23.75 (13) | 23.75 (19)
  HPA | 26.44 (24) | 21.92 (10) | 22.53 (22)

21. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Severe TEAEs and Related TEAEs: Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were are any untoward medical incidence in a participant during administered study intervention, whether or not these events are related to study intervention. Severe TEAEs were defined as type of AE that interrupted usual activities of daily life (ADL), or significantly affects clinical status, or may require intensive therapeutic intervention. Related TEAEs are defined as all TEAEs considered by the investigator to have at least a 'possible' relationship with the study intervention.
Time Frame: From start of treatment up to 28 to 35 days post last dose of study intervention (approximately 52 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and received at least 1 dose of study intervention. Participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo for CTB 400 mg + AVP 900 mg (Part-1): Healthy participants were administered a single oral dose of placebo for CTB 400 mg along with a single oral dose of AVP 900 mg in any of the treatment periods.
- Placebo for CTB 800 mg + AVP 1350 mg: Healthy participants were administered a single oral dose of placebo for CTB 800 mg along with a single oral dose of AVP 1350 mg in any of the treatment periods.
- Placebo for CTB 800 mg (Part-1): Healthy participants were administered a single oral dose of placebo for CTB 800 mg in any of the treatment periods.
- Placebo for CTB 1200 mg + AVP 1350 mg (Part-1): Healthy participants were administered a single oral dose of placebo for CTB 1200 mg along with a single oral dose of AVP 1350 mg in any of the treatment periods.
- Placebo for CTB 1600 mg (Part-1): Healthy participants were administered a single oral dose of placebo for CTB 1600 mg in any of the treatment periods.
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  TEAEs | 2 | 0 | 3 | 1 | 0 | 0 | 3 | 1 | 3 | 0
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related TEAEs | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0

22. Primary Outcome: Number of Participants With Withdrawals Due to TEAEs: Part 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were are any untoward medical incidence in a participant during administered study intervention, whether or not these events are related to study intervention.
Time Frame: From start of treatment up to 28 to 35 days post last dose of study intervention (approximately 52 days)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Primary Outcome: Number of Participants With Laboratory Test Abnormalities: Part 1
Description: The laboratory abnormalities with non-zero participants were reported and it included: monocytes or leukocytes (greater than [>] 1.2* upper limit of normal [ULN]), urine hemoglobin scalar (greater than or equal to [>=1]) and leukocyte esterase scalar (>=1).
Time Frame: Up to 24 hours post-dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants
  Monocytes/Leukocytes | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
  Urine Hemoglobin (Scalar) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
  Leukocyte Esterase (Scalar) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

24. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Abnormalities: Part 1
Description: Vital signs included blood pressure and pulse rate and were measured in a supine position after approximately 5 minutes of rest for the participant. Clinically significant changes in vital signs were determined by the investigator.
Time Frame: Up to 24 hours post-dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities: Part 1
Description: Twelve lead ECGs were collected using an ECG machine that automatically calculated heart rate and measured PR interval, QRS duration, QT interval, QT interval correct by Bazzette's formula (QTcB) and QT interval correct by Frederica formula QTcF. ECG abnormalities included: PR interval aggregate (millisecond [msec], maximum [max.] >=300; baseline > 200 and max. increase >= 25 percent (%); baseline > 200 and max. increase >= 25%), QRS duration aggregate (msec, max >=140; max. increase >= 50%), QT interval aggregate (msec, value > 500), QTCB interval aggregate and QTCF interval aggregate (msec, 450 < max <= 480; 480 < max. <= 500; max. > 500; 30 < max. increase <= 60; max. increase > 60).
Time Frame: Up to 24 hours post-dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Maximum Observed Concentration (Cmax) of Cis-CTB and Trans-CTB: Part 2
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6 and 8 hours post dose on Day 1 and 6; pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,16 and 24 hours post dose on Day 7
Population: Pharmacokinetic parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported for the given part of the study. Trans-CTB was measured only for CTB400 mg+AVP 1350 mg q8h arm as pre-specified in the protocol. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter
  Cis-CTB Day 1 | 14610 (21) | 22730 (26) | 17270 (11)
  Cis-CTB Day 6: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 6 | 22630 (7) | 45640 (24) | 20680 (16)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 21660 (17) | 35240 (25) | 20390 (10)
  Trans-CTB Day 1: number analyzed (Participants) | 6 | 0 | 0
  Trans-CTB Day 1 | 834.7 (17) |  |
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 1428 (12) |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 1641 (15) |  |
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 104.47, 90% CI 2-sided [84.94 to 128.50] — Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect (fed vs fasted)
Statistical Analysis 2: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 129.54, 90% CI 2-sided [119.37 to 140.58] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 101.46, 90% CI 2-sided [88.68 to 116.08] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); Trans-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric means = 86.99, 90% CI 2-sided [74.48 to 101.59] — Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect (fed vs fasted) for CTB 400 mg + AVP 1350 mg only

27. Primary Outcome: Time for Cmax (Tmax) of Cis-CTB and Trans-CTB: Part 2
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Median (Full Range); unit: Hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  Cis-CTB Day 1 | 2.54 [2.03 to 4.22] | 3.53 [2.03 to 4.03] | 2.53 [1.53 to 6.03]
  Cis-CTB Day 6: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 6 | 2.80 [2.03 to 4.03] | 3.53 [2.53 to 4.05] | 3.28 [1.05 to 6.03]
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 2.05 [1.53 to 2.53] | 2.03 [1.53 to 2.55] | 2.29 [1.53 to 3.03]
  Trans-CTB Day 1: number analyzed (Participants) | 6 | 0 | 0
  Trans-CTB Day 1 | 5.13 [4.03 to 6.08] |  |
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 3.54 [3.03 to 4.03] |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 3.54 [3.03 to 4.03] |  |

28. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Time Tau, the Dosing Interval (AUCtau) of Cis-CTB and Trans-CTB: Part 2
Description: Area under the plasma concentration time profile from time zero to time tau, the dosing interval, where tau is equal to 8 hours for three times daily (TID) dosing.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6 and 8 hours post dose on Day 1 and 6; pre-dose,0.5,1,1.5,2,2.5,3,4,6 and 8 hours post dose on Day 7
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hours per milliliter
  Cis-CTB Day 1 | 64640 (14) | 113100 (22) | 67730 (11)
  Cis-CTB Day 6: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 6 | 104200 (10) | 224300 (23) | 93590 (17)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 101900 (11) | 167600 (24) | 93660 (8)
  Trans-CTB Day 1: number analyzed (Participants) | 6 | 0 | 0
  Trans-CTB Day 1 | 4112 (13) |  |
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 8968 (11) |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 10060 (12) |  |
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 102.21, 90% CI 2-sided [88.67 to 117.80] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 133.79, 90% CI 2-sided [119.84 to 149.36] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); Cis-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 99.93, 90% CI 2-sided [90.70 to 110.10] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); Trans-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 89.17, 90% CI 2-sided [75.27 to 105.63] — [estimate comment as in outcome 26, analysis 4]

29. Primary Outcome: Dose-Normalized Cmax (Cmax[dn]) of Cis-CTB and Trans-CTB : Part 2
Description: Dose-normalized Cmax was determined as Cmax/Dose.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter per milligram
  Cis-CTB Day 1 | 36.56 (21) | 28.43 (26) | 43.22 (11)
  Cis-CTB Day 6: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 6 | 56.59 (7) | 57.06 (24) | 51.72 (16)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 54.21 (17) | 44.08 (25) | 51.00 (10)
  Trans-CTB Day 1: number analyzed (Participants) | 6 | 0 | 0
  Trans-CTB Day 1 | 2.089 (17) |  |
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 3.572 (12) |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 4.105 (15) |  |

30. Primary Outcome: Dose-Normalized AUCtau (AUCtau[dn]) of Cis-CTB and Trans-CTB: Part 2
Description: as for outcome 28
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hour/milliliter/milligram
  Cis-CTB Day 1 | 161.6 (14) | 141.6 (22) | 169.5 (11)
  Cis-CTB Day 6: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 6 | 260.4 (9) | 280.7 (23) | 234.2 (17)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 255.6 (11) | 209.8 (24) | 234.1 (8)
  Trans-CTB Day 1: number analyzed (Participants) | 6 | 0 | 0
  Trans-CTB Day 1 | 10.28 (13) |  |
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 22.45 (11) |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 25.20 (12) |  |

31. Primary Outcome: Terminal Half-Life (t1/2) of Cis-CTB and Trans-CTB on Day 7: Part 2
Description: as for outcome 8
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,16 and 24 hours post dose on Day 7
Population: Pharmacokinetic parameter analysis set. Trans-CTB was measured only for CTB400 mg+AVP 1350 mg q8h arm as pre-specified in the protocol. Trans-CTB was measured only for CTB400 mg+AVP 1350 mg q8h arm as pre-specified in the protocol. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
hours
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 3.710 (0.47011) | 3.930 (0.61106) | 3.030 (0.32668)
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 4.040 (0.84699) |  |

32. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Cis-CTB and Trans-CTB : Part 2
Description: as for outcome 9
Time Frame: as for outcome 26
Population: Pharmacokinetic parameter analysis set. Trans-CTB was measured only for CTB400 mg+AVP 1350 mg q8h arm as pre-specified in the protocol. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Liter
  Cis-CTB Day 1: number analyzed (Participants) | 2 | 1 | 4
  Cis-CTB Day 1 | 16.5 (13.7) | 15.6 (NA) — Geometric CV could not be calculated as only 1 participant was analyzed. | 15.37 (15)
  Cis-CTB Day 6: number analyzed (Participants) | 2 | 2 | 2
  Cis-CTB Day 6 | 16.5 (13.8) | 11.5 (8.95) | 14.8 (11.2)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 20.86 (22) | 26.76 (36) | 18.58 (13)
  Trans-CTB Day 1: number analyzed (Participants) | 0 | 0 | 0
  Trans-CTB Day 6: number analyzed (Participants) | 0 | 0 | 0
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 227.5 (25) |  |

33. Primary Outcome: Apparent Clearance (CL/F) of Cis-CTB and Trans-CTB: Part 2
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: as for outcome 26
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour
  Cis-CTB Day 1: number analyzed (Participants) | 2 | 1 | 4
  Cis-CTB Day 1 | 4.61 (4.45) | 4.89 (NA) — Geometric CV could not be calculated as only 1 participant was analyzed. | 5.014 (10)
  Cis-CTB Day 6: number analyzed (Participants) | 2 | 2 | 2
  Cis-CTB Day 6 | 3.844 (10) | 3.579 (23) | 4.283 (17)
  Cis-CTB Day 7: number analyzed (Participants) | 4 | 6 | 6
  Cis-CTB Day 7 | 3.914 (11) | 4.774 (24) | 4.273 (8)
  Trans-CTB Day 1: number analyzed (Participants) | 0 | 0 | 0
  Trans-CTB Day 6: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 6 | 44.85 (12) |  |
  Trans-CTB Day 7: number analyzed (Participants) | 4 | 0 | 0
  Trans-CTB Day 7 | 39.67 (12) |  |

34. Primary Outcome: Maximum Observed Concentration (Cmax) of AVP, AVI and HPA: Part 2
Description: The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: as for outcome 26
Population: Pharmacokinetic parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported for the given part of the study. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter
  AVP Day 1 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVP Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVP Day 7 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 1 | 6249 (25) | 5852 (12) | 4779 (27)
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 7940 (15) | 8676 (37) | 6159 (15)
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 8474 (12) | 7673 (20) | 5753 (12)
  HPA Day 1 | 2568 (29) | 2539 (10) | 1977 (25)
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 3216 (28) | 3432 (35) | 2643 (20)
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 3986 (24) | 3817 (21) | 2707 (15)
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 93.69, 90% CI 2-sided [78.37 to 112.02] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); AVI-CTB Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 113.07, 90% CI 2-sided [88.31 to 144.76] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 107.06, 90% CI [92.77 to 123.54] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 80.68, 90% CI 2-sided [68.32 to 95.27] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 5: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 89.92, 90% CI 2-sided [69.70 to 116.02] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 6: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 97.65, 90% CI 2-sided [84.08 to 113.41] — [estimate comment as in outcome 26, analysis 1]

35. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Time Tau, the Dosing Interval (AUCtau) of AVP, AVI and HPA: Part 2
Description: as for outcome 28
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hours per milliliter
  AVP Day 1: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 0
  AVI Day 1 | 29480 (16) | 27920 (24) | 22530 (15)
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 39570 (14) | 45130 (21) | 29920 (17)
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 38670 (16) | 38300 (19) | 25810 (9)
  HPA Day 1 | 12310 (28) | 12740 (23) | 9623 (22)
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 17910 (32) | 20020 (30) | 14190 (22)
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 21000 (22) | 20500 (22) | 13790 (16)
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 102.33, 90% CI 2-sided [90.37 to 115.87] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 117.83, 90% CI 2-sided [100.61 to 138.00] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 115.88, 90% CI 2-sided [104.12 to 128.98] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 85.27, 90% CI 2-sided [70.37 to 103.32] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 5: Comparison: CTB 800 mg + AVP 1350 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 97.69, 90% CI 2-sided [78.83 to 121.06] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 6: Comparison: CTB 400 mg + AVP 900 mg q8h (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 102.85, 90% CI 2-sided [94.80 to 111.58] — [estimate comment as in outcome 26, analysis 1]

36. Primary Outcome: Time for Cmax (Tmax) of AVP, AVI and HPA: Part 2
Description: The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Median (Full Range); unit: Hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  AVP Day 1: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 1
  AVP Day 7 |  |  | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  AVI Day 1 | 4.02 [2.50 to 6.00] | 4.00 [2.50 to 6.00] | 4.49 [1.50 to 6.02]
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 2.77 [2.00 to 4.00] | 2.50 [0.000 to 4.00] | 2.75 [1.02 to 6.00]
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 1.75 [1.00 to 3.00] | 2.00 [1.00 to 4.00] | 2.54 [1.00 to 3.00]
  HPA Day 1 | 5.02 [2.50 to 6.02] | 4.00 [2.50 to 6.00] | 4.49 [1.50 to 6.02]
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 2.52 [2.00 to 4.00] | 2.50 [0.000 to 3.00] | 2.02 [0.500 to 6.00]
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 1.75 [0.500 to 3.00] | 2.26 [1.00 to 4.00] | 2.30 [1.00 to 3.00]

37. Primary Outcome: Dose-Normalized Cmax (Cmax[dn]) of AVP, AVI and HPA: Part 2
Description: Dose-normalized Cmax was determined as Cmax/Dose. The lower limit of quantification for AVP was 1.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter per milligram
  AVP Day 1 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVP Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVP Day 7 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 1 | 6.907 (25) | 6.470 (12) | 7.927 (27)
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 8.786 (15) | 9.587 (37) | 10.21 (15)
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 9.373 (12) | 8.483 (20) | 9.544 (12)
  HPA Day 1 | 6.340 (29) | 6.270 (10) | 7.324 (25)
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 7.939 (28) | 8.471 (35) | 9.782 (20)
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 9.824 (23) | 9.430 (21) | 10.02 (15)

38. Primary Outcome: Dose-Normalized AUCtau (AUCtau[dn]) of AVP, AVI and HPA: Part 2
Description: as for outcome 28
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hour/milliliter/milligram
  AVP Day 1: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 0
  AVI Day 1 | 32.63 (16) | 30.88 (24) | 37.37 (15)
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 43.77 (14) | 49.92 (21) | 49.62 (17)
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 42.73 (16) | 42.32 (19) | 42.81 (9)
  HPA Day 1 | 30.43 (28) | 31.53 (23) | 35.63 (21)
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 44.19 (32) | 49.40 (30) | 52.59 (22)
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 51.84 (22) | 50.56 (22) | 51.08 (16)

39. Primary Outcome: Terminal Half-Life (t1/2) of AVP, AVI and HPA on Day 7: Part 2
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The lower limit of quantification for HPA was 10.0 ng/mL.
Time Frame: pre-dose,0.5,1,1.5,2,2.5,3,4,6,8,12,16 and 24 hours post dose on day 7
Population: Pharmacokinetic parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported for the given part of the study. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
hours
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 0
  AVI Day 7: number analyzed (Participants) | 3 | 6 | 6
  AVI Day 7 | 6.473 (1.0929) | 8.165 (1.3241) | 7.150 (1.8379)
  HPA Day 7: number analyzed (Participants) | 3 | 2 | 6
  HPA Day 7 | 6.270 (0.64211) | NA (NA) — Data could not be calculated as values were below limit of quantification. | 5.965 (1.1229)

40. Primary Outcome: Apparent Volume of Distribution (Vz/F) of AVP, AVI and HPA: Part 2
Description: Vz/F was calculated as Dose/(AUCinf * kel) where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The lower limit of quantification for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Liter
  AVP Day 1: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 0
  AVI Day 1: number analyzed (Participants) | 0 | 0 | 3
  AVI Day 1 |  |  | 63.23 (10)
  AVI Day 6: number analyzed (Participants) | 2 | 3 | 4
  AVI Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. | 58.04 (25) | 64.02 (22)
  AVI Day 7: number analyzed (Participants) | 3 | 6 | 6
  AVI Day 7 | 228.7 (22) | 275.1 (21) | 234.7 (18)
  HPA Day 1: number analyzed (Participants) | 0 | 0 | 2
  HPA Day 1 |  |  | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 6: number analyzed (Participants) | 1 | 0 | 1
  HPA Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. |  | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 3 | 2 | 6
  HPA Day 7 | 188.1 (24) | NA (NA) — Data could not be calculated as values were below limit of quantification. | 165.9 (9)

41. Primary Outcome: Apparent Clearance (CL/F) of AVP, AVI and HPA: Part 2
Description: CL/F was calculated as Dose/AUCinf.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2)
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour
  AVP Day 1: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0 | 0
  AVI Day 1 | 30.65 (16) | 32.38 (24) | 26.76 (15)
  AVI Day 6: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 6 | 22.86 (14) | 20.02 (21) | 20.13 (17)
  AVI Day 7: number analyzed (Participants) | 4 | 6 | 6
  AVI Day 7 | 23.41 (16) | 23.61 (19) | 23.34 (9)
  HPA Day 1 | 32.89 (28) | 31.73 (23) | 28.07 (21)
  HPA Day 6: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 6 | 22.64 (32) | 20.25 (30) | 19.02 (22)
  HPA Day 7: number analyzed (Participants) | 4 | 6 | 6
  HPA Day 7 | 19.28 (22) | 19.78 (22) | 19.59 (16)

42. Primary Outcome: Number of Participants With TEAEs, Severe TEAEs and Related TEAEs: Part 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were are any untoward medical incidence in a participant during administered study intervention, whether or not these events are related to study intervention. Severe TEAEs were defined as type of AE that interrupted usual ADL, or significantly affects clinical status, or may require intensive therapeutic intervention. Related TEAEs are defined as all TEAEs considered by the investigator to have at least a 'possible' relationship with the study intervention.
Time Frame: From start of treatment up to 28 to 35 days post last dose of study intervention (approximately 42 days)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Groups:
- CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part 2): Healthy Japanese participants were administered CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part 2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1
Participants
  TEAEs | 5 | 2 | 4 | 1 | 5 | 2 | 2 | 0 | 3 | 0
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related TEAEs | 4 | 1 | 4 | 1 | 3 | 2 | 1 | 0 | 3 | 0

43. Primary Outcome: Number of Participants With Withdrawals Due to TEAEs: Part 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any untoward medical incidence in a participant during administered study intervention, whether or not these events are related to study intervention.
Time Frame: From start of treatment up to 28 to 35 days post last dose of study intervention (approximately 42 days)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part 2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1
Participants | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

44. Primary Outcome: Number of Participants With Laboratory Test Abnormalities: Part 2
Description: The laboratory abnormalities with non-zero participants were reported and it included: neutrophils/ leukocytes (less than [<] 0.8x lower limit of normal [LLN]), eosinophils/leukocytes (>1.2x ULN), monocytes/leukocytes (>1.2x ULN), bicarbonate (>1.1x ULN), urine glucose (>=1), ketones scalar (>=1), urine hemoglobin scalar (>=1), leukocyte esterase scalar (>=1).
Time Frame: From start of treatment up to Day 7
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Groups:
- CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2: Healthy Japanese participants were administered CTB 400 mg along with AVP 1350 mg q8h in a fed state on Days 1 to 6 and in a fasted state on Day 7.
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2 | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1
Participants
  Neutrophils/leukocytes | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Eosinophils/leukocytes | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Monocytes/leukocytes | 1 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0
  Bicarbonate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urine glucose | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ketones (scalar) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine hemoglobin (scalar) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Leukocyte esterase (scalar) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

45. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Abnormalities: Part 2
Description: as for outcome 24
Time Frame: From start of treatment up to Day 7
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part 2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities: Part 2
Description: as for outcome 25
Time Frame: From start of treatment up to Day 7
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part 2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 5 | 1 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Amount Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau) of Cis-CTB, Trans-CTB, AVP, AVI and HPA: Part 2
Time Frame: anytime between 0 to 8 hours post dose on Day 6
Population: Pharmacokinetic analysis set. Data was planned to be analyzed for CTB 400 mg + AVP 1350 mg arm only as pre-specified in the protocol. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2)
Number analyzed (Participants) | 6
Milligrams
  Cis CTB Day 6: number analyzed (Participants) | 5
  Cis CTB Day 6 | 181.8 (98)
  Trans CTB Day 6: number analyzed (Participants) | 5
  Trans CTB Day 6 | 48.23 (54)
  AVP Day 6: number analyzed (Participants) | 0
  AVI Day 6: number analyzed (Participants) | 5
  AVI Day 6 | 295.6 (101)
  HPA Day 6: number analyzed (Participants) | 5
  HPA Day 6 | 22.01 (51)

48. Secondary Outcome: Percent of Dose Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau%) of Cis-CTB, Trans-CTB, AVP, AVI and HPA: Part 2
Description: Aetau% was calculated as 100*Aetau/Dose.
Time Frame: anytime between 0 to 8 hours post dose on Day 6
Population: as for outcome 47
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose excreted
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2)
Number analyzed (Participants) | 6
Percentage of dose excreted
  Cis CTB Day 6: number analyzed (Participants) | 5
  Cis CTB Day 6 | 45.40 (98)
  Trans CTB Day 6: number analyzed (Participants) | 5
  Trans CTB Day 6 | 12.08 (55)
  AVP Day 6: number analyzed (Participants) | 0
  AVI Day 6: number analyzed (Participants) | 5
  AVI Day 6 | 32.68 (101)
  HPA Day 6: number analyzed (Participants) | 5
  HPA Day 6 | 5.434 (51)

49. Secondary Outcome: Renal Clearance (CLr) of Cis-CTB, Trans-CTBa, AVP, AVI and HPA: Part 2
Description: Aetau% was calculated as 100*Aetau/Dose.
Time Frame: anytime between 0 to 8 hours post dose on Day 6
Population: as for outcome 47
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Part-2)
Number analyzed (Participants) | 6
Liter per hour
  Cis CTB Day 6: number analyzed (Participants) | 4
  Cis CTB Day 6 | 2.501 (27)
  Trans CTB Day 6: number analyzed (Participants) | 4
  Trans CTB Day 6 | 6.657 (27)
  AVP Day 6: number analyzed (Participants) | 0
  AVI Day 6: number analyzed (Participants) | 4
  AVI Day 6 | 10.61 (34)
  HPA Day 6: number analyzed (Participants) | 4
  HPA Day 6 | 1.390 (22)

50. Secondary Outcome: Maximum Observed Concentration (Cmax) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Nanogram per milliliter
  Cis CTB Day 1 | 13660 (35) | 19540 (16)
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 22080 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 21330 (14) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 5167 (49) | 6858 (24)
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 7677 (24) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 7279 (15) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 2248 (45) | 3341 (33)
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 3380 (14) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 3708 (8) | NA (NA) — Data could not be calculated as values were below limit of quantification.
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 105.47, 90% CI 2-sided [86.64 to 128.39] — Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect (Japanese participants fed vs fasted and Chinese participants fed vs fasted)
Statistical Analysis 2: Comparison: CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 134.24, 90% CI [51.81 to 347.81] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 91.17, 90% CI [79.54 to 104.51] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 115.26, 90% CI 2-sided [71.46 to 185.90] — [estimate comment as in outcome 50, analysis 1]

51. Secondary Outcome: Time for Cmax (Tmax) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Median (Full Range); unit: Hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Hours
  Cis CTB Day 1 | 4.03 [4.03 to 6.03] | 3.05 [2.57 to 4.05]
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 3.03 [2.53 to 4.03] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 2.03 [1.53 to 3.03] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 6.00 [1.50 to 6.00] | 3.02 [3.00 to 6.02]
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 4.00 [2.50 to 6.02] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 1.50 [1.00 to 2.50] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 6.00 [1.00 to 6.00] | 4.00 [2.50 to 6.02]
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 2.50 [2.00 to 6.02] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 2.00 [0.500 to 3.00] | NA [NA to NA] — Data could not be calculated as values were below limit of quantification.

52. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Time Tau, the Dosing Interval (AUCtau) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: Area under the plasma concentration time profile from time zero to time tau, the dosing interval, where tau is equal to 8 hours for TID dosing. The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours per milliliter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Nanogram*hours per milliliter
  Cis CTB Day 1 | 52630 (20) | 84790 (17)
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 92920 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 90270 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 22240 (33) | 32650 (32)
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 38010 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 33100 (8) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 10400 (35) | 16670 (35)
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 19160 (7) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 18890 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
Statistical Analysis 1: Comparison: CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 114.83, 90% CI 2-sided [101.10 to 130.43] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 2: Comparison: CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2); AVI- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 140.44, 90% CI 2-sided [104.17 to 189.34] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 3: Comparison: CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric mean = 101.46, 90% CI [90.79 to 113.39] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 4: Comparison: CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2); HPA- Day 6 versus Day 7; Test type: Other; Ratio of adjusted geometric means = 123.20, 90% CI 2-sided [110.25 to 137.67] — Model is a mixed effect model with treatment as a fixed effect and participant as a random effect (Japanese participants fed vs fasted and Chinese participants fed vs fasted)

53. Secondary Outcome: Dose-Normalized Cmax (Cmax[dn]) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: Dose-normalized Cmax was determined as Cmax/Dose. The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Nanogram per milliliter per milligram
  Cis CTB Day 1 | 34.16 (35) | 48.90 (16)
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 55.21 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 53.35 (14) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 5.714 (49) | 7.582 (24)
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 8.483 (24) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 8.046 (15) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 5.549 (45) | 8.249 (33)
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 8.339 (14) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 9.145 (8) | NA (NA) — Data could not be calculated as values were below limit of quantification.

54. Secondary Outcome: Dose-Normalized AUCtau (AUCtau[dn]) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: as for outcome 52
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Nanogram*hour/milliliter/milligram
  Cis CTB Day 1 | 131.5 (19) | 212.0 (17)
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 232.3 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 225.9 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 24.62 (33) | 36.10 (32)
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 42.01 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 36.59 (8) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 25.70 (35) | 41.23 (35)
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 47.29 (7) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 46.65 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.

55. Secondary Outcome: Terminal Half-Life (t1/2) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: Pharmacokinetic analysis set. It was planned to report data for CTB 400 mg + AVP 1350 mg only. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Hours
  Cis CTB Day 1: number analyzed (Participants) | 0 | 0
  Cis CTB Day 6: number analyzed (Participants) | 0 | 0
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 2.788 (0.80670) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1: number analyzed (Participants) | 0 | 0
  AVI Day 6: number analyzed (Participants) | 0 | 0
  AVI Day 7: number analyzed (Participants) | 5 | 1
  AVI Day 7 | 5.734 (2.6304) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1: number analyzed (Participants) | 0 | 0
  HPA Day 6: number analyzed (Participants) | 0 | 0
  HPA Day 7: number analyzed (Participants) | 5 | 1
  HPA Day 7 | 5.290 (1.7122) | NA (NA) — Data could not be calculated as values were below limit of quantification.

56. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: Vz/F was calculated as Dose/(AUCinf * kel) where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Liter
  Cis CTB Day 1: number analyzed (Participants) | 0 | 1
  Cis CTB Day 1 |  | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 6: number analyzed (Participants) | 4 | 0
  Cis CTB Day 6 | 12.82 (8) |
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 17.33 (31) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1: number analyzed (Participants) | 0 | 0
  AVI Day 6: number analyzed (Participants) | 1 | 1
  AVI Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 1
  AVI Day 7 | 207.9 (43) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1: number analyzed (Participants) | 0 | 0
  HPA Day 6: number analyzed (Participants) | 1 | 1
  HPA Day 6 | NA (NA) — Data could not be calculated as values were below limit of quantification. | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 1
  HPA Day 7 | 156.0 (44) | NA (NA) — Data could not be calculated as values were below limit of quantification.

57. Secondary Outcome: Apparent Clearance (CL/F) of Cis-CTB, AVP, AVI and HPA in Japanese and Chinese Cohorts: Part 2
Description: CL/F was calculated as Dose/AUCinf. The lower limit of quantification for cis-CTB was 100.0 ng/mL, and for AVI and HPA was 10.0 ng/mL.
Time Frame: as for outcome 26
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
Number analyzed (Participants) | 5 | 3
Liter/hour
  Cis CTB Day 1: number analyzed (Participants) | 0 | 1
  Cis CTB Day 1 |  | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 6: number analyzed (Participants) | 5 | 2
  Cis CTB Day 6 | 4.303 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  Cis CTB Day 7: number analyzed (Participants) | 5 | 2
  Cis CTB Day 7 | 4.428 (9) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVP Day 1: number analyzed (Participants) | 0 | 0
  AVP Day 6: number analyzed (Participants) | 0 | 0
  AVP Day 7: number analyzed (Participants) | 0 | 0
  AVI Day 1 | 40.66 (33) | 27.69 (32)
  AVI Day 6: number analyzed (Participants) | 5 | 2
  AVI Day 6 | 23.80 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  AVI Day 7: number analyzed (Participants) | 5 | 2
  AVI Day 7 | 27.33 (8) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 1 | 38.94 (35) | 24.26 (35)
  HPA Day 6: number analyzed (Participants) | 5 | 2
  HPA Day 6 | 21.12 (7) | NA (NA) — Data could not be calculated as values were below limit of quantification.
  HPA Day 7: number analyzed (Participants) | 5 | 2
  HPA Day 7 | 21.42 (11) | NA (NA) — Data could not be calculated as values were below limit of quantification.

ADVERSE EVENTS:
Time Frame: From start of treatment up to 28 to 35 days post last dose of study intervention (approximately 52 days for part 1 and 42 days for part 2)
Groups:
- Placebo for CTB 800 mg + AVP 1350 mg (Part-1): Healthy participants were administered a single oral dose of placebo for CTB 800 mg along with a single oral dose of AVP 1350 mg in any of the treatment periods.
Arm/Group | CTB 400 mg + AVP 900 mg (Part-1) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) | CTB 800 mg + AVP 1350 mg (Part-1) | Placebo for CTB 800 mg + AVP 1350 mg (Part-1) | CTB 800 mg (Part-1) | Placebo for CTB 800 mg (Part-1) | CTB 1200 mg + AVP 1350 mg (Part-1) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) | CTB 1600 mg (Part-1) | Placebo for CTB 1600 mg (Part-1) | CTB 400 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) | CTB 400 mg + AVP 900 mg q8h (Part-2) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/5 | 0/1 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/5 | 0/1 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/6 | 0/2 | 3/6 | 1/2 | 0/6 | 0/2 | 3/6 | 1/2 | 3/6 | 0/2 | 5/6 | 2/2 | 4/6 | 1/2 | 5/6 | 2/2 | 2/5 | 0/1 | 3/3 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CTB 400 mg + AVP 900 mg (Part-1) (N=6) | Placebo for CTB 400 mg + AVP 900 mg (Part-1) (N=2) | CTB 800 mg + AVP 1350 mg (Part-1) (N=6) | Placebo for CTB 800 mg + AVP 1350 mg (Part-1) (N=2) | CTB 800 mg (Part-1) (N=6) | Placebo for CTB 800 mg (Part-1) (N=2) | CTB 1200 mg + AVP 1350 mg (Part-1) (N=6) | Placebo for CTB 1200 mg + AVP 1350 mg (Part-1) (N=2) | CTB 1600 mg (Part-1) (N=6) | Placebo for CTB 1600 mg (Part-1) (N=2) | CTB 400 mg + AVP 1350 mg q8h (Part-2) (N=6) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Part-2) (N=2) | CTB 800 mg + AVP 1350 mg q8h (Part-2) (N=6) | Placebo for CTB 800 mg + AVP 1350 mg q8h (Part-2) (N=2) | CTB 400 mg + AVP 900 mg q8h (Part-2) (N=6) | Placebo for CTB 400 mg + AVP 900 mg q8h (Part-2) (N=2) | CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) (N=5) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Japanese) (Part-2) (N=1) | CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) (N=3) | Placebo for CTB 400 mg + AVP 1350 mg q8h (Chinese) (Part-2) (N=1)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT05554237/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT05554237/SAP_001.pdf